CLINICAL TRIAL: NCT06641466
Title: AN INTERVENTIONAL EFFICACY AND SAFETY, PHASE 3, DOUBLE-BLIND, PARALLEL GROUP STUDY TO INVESTIGATE INTERMITTENT PREVENTION OF MENSTRUAL MIGRAINE WITH RIMEGEPANT COMPARED WITH PLACEBO IN WOMEN PARTICIPANTS 18 TO 45 YEARS OF AGE
Brief Title: A Study to Learn About the Study Medicine Called Rimegepant in Women When Used for Intermittent Prevention of Menstrual Migraine
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C4951063; NCT06641466 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Menstrual Migraine
MeSH Terms: interventions — rimegepant sulfate; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Rimegepant 75 mg Orally Disintegrating Tablet (ODT) 7-Day Dosing (Experimental)
  Interventions: Drug: Rimegepant
- Rimegepant 75 mg Orally Disintegrating Tablet (ODT) Acute Treatment Dosing (Experimental)
  Interventions: Drug: Rimegepant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator
- Standard of Care (Active Comparator)
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Rimegepant — Rimegepant 75 mg ODT for 7 days
  Arms: Rimegepant 75 mg Orally Disintegrating Tablet (ODT) 7-Day Dosing
Drug: Placebo Comparator — Matching placebo oral disintegrating tablets for 7 days
  Arms: Placebo
Drug: Standard of Care — Standard of care for acute treatment as needed
  Arms: Standard of Care
Drug: Rimegepant — Rimegepant 75 mg ODT for acute treatment as needed
  Arms: Rimegepant 75 mg Orally Disintegrating Tablet (ODT) Acute Treatment Dosing

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rimegepant when administered during the peri-menstrual period (PMP) for intermittent prevention of migraine in women who experience menstrual migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has regular menstrual cycles ≥24 days and ≤34 days
2. A minimum 1-year history of migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition
3. A history of menstrual migraine attacks of at least 3 months
4. Participant reported history of experiencing at least 1 migraine attack during the perimenstrual period in at least 2 out of 3 menstrual cycles immediately prior to screening.
5. If the participant is receiving a permitted background continuous prophylactic migraine medication, the medication dose must be stable for at least 3 months prior to the Screening visit and, the dose is not expected to change during the course of the study

Exclusion Criteria:

1. Greater than 6 migraine days per month that are outside of the perimenstrual period in the 3 months prior to Screening
2. A diagnosis of chronic migraine or a history of more than 14 headache days per month on average, in the 3 months prior to Screening
3. History of retinal migraine, basilar migraine or hemiplegic migraine
4. Current diagnosis of schizophrenia, bipolar, or borderline personality disorder
5. Other pain syndromes (eg, fibromyalgia, complex regional pain syndrome), or significant neurological disorders (other than migraine), or other medical conditions (including endocrine and gynecological eg, severe dysmenorrhea

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 723 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-11-29 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Mean change from the Observation Period in number of migraine days per 5-day perimenstrual period across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from Observation Period in the number of migraine days per the 5-day perimenstrual period

SECONDARY OUTCOMES:
Mean change from the Observation Period in number of headache days per 5-day perimenstrual period across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from the Observation Period in number of headache days per 5-day perimenstrual period
Percentage of participants with ≥50% reduction from the Observation Period in number of migraine days per 5-day perimenstrual period across each cycle of the Double-Blind Treatment Phase (50% responder) | 5 months (5 menstrual cycles)
  Patients with ≥50% reduction from the Observation Period in number of migraine days per 5-day perimenstrual period
Mean change from the Observation Period in number of acute migraine medication days per 5-day perimenstrual period across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from the Observation Period in number of acute migraine medication days per 5-day perimenstrual period
Mean change from the Observation Period in number of acute migraine-specific medication days per 5-day perimenstrual period across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from the Observation Period in number of acute migraine specific medication days per 5-day perimenstrual period
Mean change from the Observation Period in number of migraine days with moderate-severe functional disability per 5-day perimenstrual period across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from the Observation Period in number of migraine days with moderate-severe functional disability per 5-day perimenstrual period
Mean change from the Observation Period in number of moderate-severe headache days per 5-day perimenstrual period across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from the Observation Period in number of moderate-severe headache days per 5-day perimenstrual period
Mean change from the Observation Period in number of moderate-severe migraine days per 5-day perimenstrual period across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from the Observation Phase in number of moderate-severe migraine days per 5-day perimenstrual period
Mean change from baseline in the MiCOAS Cognition score at postdosing (ie, 1 day after the 7-day dosing period) across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from baseline in the MiCOAS Cognition score at post-dosing across each cycle
Mean change from the Observation Period in monthly migraine days (per cycle, normalized to 28-days) across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from the Observation Phase in monthly migraine days
Mean change from the Observation Period in monthly headache days (per cycle, normalized to 28-days) across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from the Observation Phase in monthly headache days
Mean change from the Observation Phase in monthly acute migraine-specific medication days (per cycle, normalized to 28-days) across each cycle of the Double-Blind Treatment Phase | 5 months (5 menstrual cycles)
  Change from the Observation Phase in monthly acute migraine-specific medication days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (114):
- United States (31):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Specialty Building, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Hope Clinical Research, Inc., Canoga Park, California
  - Axiom Research, Colton, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - VIN - Aventura, Aventura, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Urban Family Practice Associates, Marietta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - St Luke's Clinic - Neurology, Meridian, Idaho
  - Alliance for Multispecialty Research - Medisphere Medical Research Center, Evansville, Indiana
  - Michigan Headache & Neurological Institute, Ann Arbor, Michigan
  - Clinvest Headlands Llc, Springfield, Missouri
  - St. Charles Clinical Research, Weldon Spring, Missouri
  - McGill Family Practice, Papillion, Nebraska
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Rochester Clinical Research, LLC, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - Thomas Jefferson University, Jefferson Headache Center, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - AMR Clinical, Knoxville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - ChronicleBio, West Valley City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - MedStar Health Neurology/MedStar Georgetown Headache Center, McLean, Virginia
- Argentina (3):
  - IDIM - Instituto de Investigaciones Metabólicas, Ciudad de Buenos Aires, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires, Buenos Aires F.D.
  - Sanatorio del Sur, San Miguel de Tucumán, Tucumán Province
- Canada (7):
  - CaRe Clinic, Red Deer, Alberta
  - OCT Research ULC, Kelowna, British Columbia
  - Centre for Neurology Studies, Surrey, British Columbia
  - Centricity Research Halifax Multispecialty, Halifax, Nova Scotia
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Centre de Recherche Saint-Louis inc., Lévis, Quebec
- China (10):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shaanxi provincial people's hospital, Xi'an, Shaanxi
  - Xianyang Hospital of Yan'an University, Xianyang, Shaanxi
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Qingdao Central Hospital, University of Health and Rehabilitation Sciences, Qingdao
  - Shanghai East Hospital, Shanghai
- Denmark (2):
  - Rigshospitalet, Glostrup, Glostrup Municipality
  - Region Midtjylland, Regionshospitalet Viborg, Viborg
- Germany (4):
  - Klinische Forschung Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Charité Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - FutureMeds GmbH, Berlin
  - Neurologie Berlin, Berlin
- India (6):
  - Lalitha Super Specialities Hospital Pvt Ltd, Guntur, Andhra Pradesh
  - Marengo CIMS Hospital, Ahmedabad, Ahmedabad, Gujarat
  - Mallikatta Neuro Centre, Mangaluru, Karnataka
  - Getwell Hospital and Research Institute, Nagpur, Maharashtra
  - Chopda Medicare & Research Centre Pvt. Ltd: Magnum Heart Institute, Nashik, Maharashtra
  - Jawahar Lal Nehru Medical College, Ajmer, Rajasthan
- Italy (6):
  - Ospedale Civile SS. Nicola e Filippo Avezzano Pronto Soccorso, Avezzano, L'aquila
  - Ospedale Bellaria- Azienda USL di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - Fondazione Istituto Neurologico C. Mondino, Pavia
  - IRCCS San Raffaele Roma, Roma
- Japan (7):
  - Konan Medical Center, Kobe, Hyōgo
  - Tatsuoka Neurology Clinic, Kyoto-shi Shimogyo-ku, Kyoto
  - Sendai Headache and Neurology Clinic, Sendai, Miyagi
  - Tokyo Headache Clinic, Shibuya-ku, Tokyo
  - Nagaseki Headache Clinic, Kai, Yamanashi
  - Tanaka Neurosurgery&Headache Clinic, Kagoshima
  - Tanaka Neurosurgical Clinic, Kagoshima
- Mexico (7):
  - Centro de Investigación Médico Biológica y Terapia Avanzada, Guadalajara, Jalisco
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Medical Care and Research SA de CV, Mérida, Yucatán
  - San Peregrino Unidad de Investigación, Aguascalientes
  - Operadora Unidad de Investigación en Salud de Chihuahua, Chihuahua City
  - PCR Cuautitlán Izcalli, Cuautitlán Izcalli
  - Clinical Research Institute S.C., Tlalnepantla
- Netherlands (3):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Isala Klinieken Stichting, Zwolle, Overijssel
  - Leids Universitair Medisch Centrum (LUMC), Leiden, South Holland
- Poland (7):
  - Instytut Zdrowia Dr Boczarska Jedynak, Oświęcim, Lesser Poland Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny, Wroclaw, Lower Silesian Voivodeship
  - NZOZ Neuromed M.i M. Nastaj, Lublin, Lublin Voivodeship
  - Indywidualna Praktyka Lekarska Dr Hab. Med. Anna Szczepanska-Szerej, Lublin, Lublin Voivodeship
  - FutureMeds Warszawa Centrum, Warsaw, Masovian Voivodeship
  - Dr Sękowska Leczenie Bólu, Warsaw, Masovian Voivodeship
  - Silmedic, Katowice, Silesian Voivodeship
- South Korea (5):
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Kyǒnggi-do
  - Ewha Womans University Seoul Hospital, Gangseo-gu, Seoul-teukbyeolsi [seoul]
  - Nowon Eulji Medical Center, Eulji University, Seoul, Seoul-teukbyeolsi [seoul]
  - Kangbuk Samsung Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (8):
  - Hospital Clínic de Barcelona, Barcelona, Barcelona [barcelona]
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - FutureMeds Spain Cádiz, Chiclana de la Frontera, Cádiz
  - Hospital La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- United Kingdom (8):
  - West Walk Surgery, Bristol, Bristol, CITY of
  - Bioluminux, Milton Keynes, Buckinghamshire
  - Hull University Teaching Hospitals NHS Trust, Hull, EAST Yorkshire
  - Re:Cognition Health - London, London, England
  - The Walton Centre NHS Foundation Trust, Liverpool, Merseyside
  - Panthera Clinic - York, York, North Yorkshire
  - Panthera Biopartners - Glasgow, Glasgow, Scotland
  - Panthera Biopartners - Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4951063